CLINICAL TRIAL: NCT00383617
Title: Performance of Referral Recommendations in Patients With Chronic Back Pain and Suspected Axial Spondyloarthritis
Brief Title: Referral Recommendations for Axial Spondyloarthritis
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, J. Sieper, Prof., Charite University, Berlin, Germany
Other Study IDs: Antragsnummer : EA4/058/05
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Spondyloarthropathy; Ankylosing Spondylitis; Spondyloarthritis
Keywords: pre-radiographic; screening; early diagnosis
MeSH Terms: conditions — Spondylarthropathies; Spondylitis, Ankylosing; Spondylarthritis; Disease

SUMMARY:
The purpose of this study is to determine which of the proposed screening parameters or which combination of screening parameters perform best in daily clinical practice for making the diagnosis of axial Spondyloarthritis (SpA)in patients with chronic low back pain.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) and its early form accounts for up to 5% of all patients with chronic back pain. Shortening the delay of 5-10 years between first symptoms and making a diagnosis of AS has become a challenge especially because effective treatments have become available. Easy to apply referral parameters for physicians in primary care may contribute to make the diagnosis earlier.

Methods: Orthopedists and primary care physicians were offered to refer patients with i) chronic low back pain (duration >3 months) and ii) onset of back pain at an age < 45 years to a specialized rheumatology outpatient clinic for further diagnostic work-up if at least one of the following screening parameters was present: 1) inflammatory back pain (IBP), 2) positive HLA-B27, 3) sacroiliitis as detected by imaging. The final diagnosis was made according to expert opinion.

It was analyzed, which parameters or combination of parameters performed best in making a diagnosis of axial SpA.

ELIGIBILITY:
Inclusion Criteria:

* chronic back pain with a duration of more than 3 months
* onset of back pain before age of 45 years

Exclusion Criteria:

* age younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Sieper, MD, Principal Investigator — Department of Rheumatology, Medical Clinic I, Charité University Medicine Berlin, Campus Benjamin Franklin, Berlin, Germany
Locations (1):
- Department of Rheumatology, Medical Clinic I, Charite Campus Benjamin Franklin, Hindenburgdamm 30, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Rudwaleit M, Khan MA, Sieper J. The challenge of diagnosis and classification in early ankylosing spondylitis: do we need new criteria? Arthritis Rheum. 2005 Apr;52(4):1000-8. doi: 10.1002/art.20990. No abstract available. PMID 15818678
- [Background] Sieper J, Rudwaleit M. Early referral recommendations for ankylosing spondylitis (including pre-radiographic and radiographic forms) in primary care. Ann Rheum Dis. 2005 May;64(5):659-63. doi: 10.1136/ard.2004.028753. Epub 2004 Nov 4. PMID 15528281